CLINICAL TRIAL: NCT00549484
Title: Thrombopoietin Levels Following Platelet Transfusion in Neonates With Thrombocytopenia
Brief Title: Thrombopoietin Levels and Platelet Transfusion in Neonates
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: T. Alex Kline, Christiana Hospital
Other Study IDs: CCC#23049
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Thrombocytopenia
Keywords: Thrombocytopenia; Thrombopoietin; Platelet Transfusion; Platelet Factor 4
MeSH Terms: conditions — Thrombocytopenia; Jacobs syndrome

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected pre and post platelet transfusion. Samples included platelet count, thrombopoietin, and platelet factor 4.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 10 mL/kg platelet transfusion
- 2: 15 mL / kg platelet transfusion

SUMMARY:
Infants who have low platelets and who require a platelet transfusion are included in this study. Platelet transfusions are routinely given to infants when their platelet count falls below a certain level. The study will look at the amount of platelets transfused. The purpose of the study is to evaluate the effect of platelet transfusions on the level of a protein (thrombopoietin) which is known to help control platelet production.

DETAILED DESCRIPTION:
Thrombocytopenia, defined as a platelet count < 150,000/mm3, is a very common hematologic problem in the neonatal period. Multiple etiologies are known to be associated with thrombocytopenia in neonates. Thrombopoietin (TPO) is known to be the central regulator of megakaryocyte and platelet production in adults and infants. However, the role of TPO in neonatal platelet regulation is not well understood. TPO levels have been shown to be higher in neonates with thrombocytopenia, with a decrease in TPO after resolution of the thrombocytopenia. The response of TPO levels in neonates after platelet transfusion has never been studied. In addition, the optimal volume of platelet transfusions has never been studied in neonates. This study will evaluate the response to 2 different volumes of platelet transfusion.

We hypothesize that a decrease in plasma TPO levels will be seen following a platelet transfusion in a population of neonates with thrombocytopenia. We also hypothesize that a platelet transfusion of 15 mL/kg will result in a greater rise in platelet count than a transfusion pf 10 mL/kg of platelets.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with thrombocytopenia
* Decision made by medical team to transfuse with platelets

Exclusion Criteria:

* Infants with major congenital malformations

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants who require platelet transfusion
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2003-05; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Reduction in TPO levels following platelet transfusion | Within 36 hours of transfusion

SECONDARY OUTCOMES:
Platelet rise following platelet transfusion in 10 mL/kg versus 15 mL/kg. | Within 36 hours after platelet transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Alex Kline, MD, Principal Investigator — Christiana Hospital; David A. Paul, MD, Principal Investigator — Christiana Hospital
Locations (1):
- Christiana Hospital, Newark, Delaware, United States